CLINICAL TRIAL: NCT07252024
Title: Nurse-Led Bispectral Index (BIS)-Guided Sedation Protocol and Its Impact on Clinical Outcomes in Mechanically Ventilated Pediatric Intensive Care Patients: A Prospective, Randomized Controlled Trial
Brief Title: Nurse-Led BIS-Guided Sedation Protocol in Pediatric Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Hasan ağın, Prof.Dr, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 02024/GOA-92
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Nurse's Role; Bispectral Index; Pediatric Sedation

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, randomized controlled trial comparing a nurse-led BIS-guided sedation protocol with standard sedation management in mechanically ventilated pediatric patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS-Guided Nurse-Led Sedation Protocol (Experimental): Patients in this arm will receive sedation management guided by a nurse-led protocol using Bispectral Index (BIS) monitoring. Nurses titrate sedative medications according to BIS targets (light sedation: 60-80; deep sedation: 45-60) and Sedation Behavioral Scale (SBS) scores, under physician supervision. The protocol includes standardized electrode placement, artifact management, and stepwise titration of midazolam, ketamine, dexmedetomidine, or fentanyl according to predefined algorithms.
  Interventions: Behavioral: BIS-Guided Sedation Protocol
- Standard Sedation Protocol (No Intervention): Patients in this arm receive routine sedation management according to the existing standard sedation protocol. Clinicians titrate sedative medications based on clinical assessment and SBS scores without using BIS-guided titration. BIS monitoring is available but not used for sedation adjustment.

INTERVENTIONS:
Behavioral: BIS-Guided Sedation Protocol — A structured sedation management protocol guided by Bispectral Index (BIS) monitoring and implemented by trained PICU nurses. The protocol includes BIS target ranges (light sedation 60-80; deep sedation 45-60), artifact recognition, standardized electrode placement, and stepwise titration of midazolam, ketamine, dexmedetomidine, or fentanyl according to predefined algorithms under physician supervision.
  Arms: BIS-Guided Nurse-Led Sedation Protocol

SUMMARY:
Pediatric intensive care sedation is traditionally based on subjective clinical scales. Bispectral Index (BIS) monitoring provides an objective EEG-based assessment of sedation depth. This prospective, two-center randomized controlled trial evaluates whether a nurse-led BIS-guided sedation protocol can reduce excessive or inadequate sedation, sedative medication exposure, withdrawal symptoms, and PICU length of stay in mechanically ventilated children.

DETAILED DESCRIPTION:
This prospective, randomized (1:1) controlled trial was conducted in two tertiary PICUs in Turkey, including mechanically ventilated children aged 1 month to 18 years requiring continuous sedation. Patients were randomly assigned to:

Intervention Group: Nurse-led sedation titration using BIS values (target: light sedation 60-80, deep sedation 45-60) combined with SBS scores under physician supervision. Nurses received structured theoretical and practical training before trial initiation.

Control Group: Standard sedation protocol based solely on clinical sedation assessment without BIS-guided titration (BIS monitoring available but not used for titration).

Primary Outcome:

Percentage and duration of time spent outside the target BIS range

Total sedative medication dose (mg/kg/day equivalents)

Secondary Outcomes:

PICU length of stay

Mechanical ventilation duration

Withdrawal symptoms (WAT-1 score)

Results showed significantly reduced BIS out-of-target time, lower sedative drug exposure (midazolam, ketamine, dexmedetomidine), reduced withdrawal scores, and shorter PICU stay in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 18 years
* Receiving invasive mechanical ventilation
* Expected to require sedation for ≥24 hours
* Hemodynamically stable at enrollment
* BIS monitoring electrode placement feasible

Exclusion Criteria:

* Use of neuromuscular blocking agents at enrollment
* Mechanical ventilation expected to last <24 hours
* Severe hemodynamic instability requiring escalating vasoactive support
* Known neurological disorders that prevent reliable BIS interpretation (e.g., severe encephalopathy, epileptic burst suppression)
* Facial burns or skin conditions preventing BIS electrode placement
* Decision for palliative/comfort care only

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Time Spent Outside BIS Target Range | First 72 hours of mechanical ventilation
  otal duration (in hours) during which BIS values remain outside the predefined sedation targets (light sedation: 60-80; deep sedation: 45-60). This measure reflects adequacy of sedation and protocol effectiveness.
Cumulative Midazolam Dose | Up to 28 days or until extubation
  otal midazolam dose administered (mg/kg) during mechanical ventilation.
Cumulative Ketamine Dose | Up to 28 days or until extubation
  Total ketamine dose administered (mcg/kg) during mechanical ventilation.
Cumulative Dexmedetomidine Dose | Up to 28 days or until extubation
  Total dexmedetomidine dose administered (mcg/kg) during mechanical ventilation.

SECONDARY OUTCOMES:
Withdrawal Severity (WAT-1 Score) | First 7 days of PICU stay
  Mean and peak WAT-1 scores assessed to determine iatrogenic withdrawal severity.
PICU Length of Stay | Up to 28 days
  Total number of days from PICU admission to PICU discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Prof.Dr., Principal Investigator — Dr. Behcet Uz Children's Hospital
Locations (1):
- Behcet Uz Children's Hospital - Pediatric Intensive Care Unit, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy and institutional policy.